CLINICAL TRIAL: NCT07400731
Title: Multicenter Study of Safety and Effectiveness of Auricular Muscle Zone Stimulation With the EarStim Novel Device for Parkinson's Disease
Brief Title: Short and Long-term Responses of PD Symptoms to Earstim
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stoparkinson Healthcare Systems LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STP-PD-006
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: parkinson disease; intrinsic auricular muscle zone stimulation; IAMZ
MeSH Terms: conditions — Parkinson Disease | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Period A of the study will be double-blind, randomized, sham-controlled. Participant and investigator will be blinded.
  Period B will be open label and SOC-controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active arm (Period A) (Experimental): Patients in the active arm in Period A will wear the investigational EarStim System
  Interventions: Device: EarStim; Device: EarStim + Standard of care (SOC)
- Sham arm (Period A) (Sham Comparator): Patients in the sham arm in Period A will wear an identical device with no active stimulation.
  Interventions: Device: Sham device; Other: Standard of Care (SOC)

INTERVENTIONS:
Device: EarStim — Patients in the active arm in Period A will wear the investigational EarStim System
  Arms: Active arm (Period A)
Device: Sham device — Patients in the sham arm in Period A will wear an identical device with no active stimulation, programmed in similar manner as the EarStim system
  Arms: Sham arm (Period A)
Device: EarStim + Standard of care (SOC) — Participants in the active arm in Period A who are responders to stimulation (based on reduction in MDS-UPDRS III scores) will proceed to Period B, which takes place in a home setting.
  In Period B, these responders will be assigned to "EarStim + SOC" group. They will be instructed to continue their oral dopaminergic medications as usual, and in addition, to use EarStim stimulation at home at the time of their medication intake.
  Arms: Active arm (Period A)
Other: Standard of Care (SOC) — Participants from the sham arm of Period A will be assigned to the "SOC" group and will continue their oral dopaminergic medications as usual, without any EarStim stimulation.
  Arms: Sham arm (Period A)

SUMMARY:
This is a prospective, multicenter, randomized, two-period study designed to evaluate the safety and effectiveness of the EarStim System for intermittent relief of motor symptoms in patients with Parkinson's disease experiencing wearing-off phenomena. Adult patients with moderate to severe Parkinson's disease (MDS-UPDRS Part III score ≥33) receiving oral dopaminergic therapy will be enrolled. Period A is a randomized, double-blind, sham-controlled phase conducted in a clinical setting. Period B is an unblinded, standard-of-care-controlled phase evaluating the effectiveness of the EarStim System during home use over 90 days.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disorder, affecting approximately 0.3% of the general population and up to 3% of individuals over 65. It is characterized by cardinal motor symptoms such as bradykinesia, rigidity, tremor, and postural instability. While levodopa remains the gold-standard treatment, long-term use often leads to motor complications, including fluctuations between "ON" and "OFF" states. Deep brain stimulation of the subthalamic nucleus is an effective intervention for motor symptoms and medication-induced complications; however, axial symptoms such as postural instability and gait disturbances remain resistant to treatment. Alternative approaches, including peripheral nerve stimulation, have been explored to modulate motor control regions of the brain, offering potential benefits for PD symptom management.

The EarStim System, developed by Stoparkinson Healthcare Systems, is a wearable, non-invasive electro-stimulator designed to target intrinsic auricular muscle zones (IAMZ). These zones are innervated by the trigeminal, facial, vagus, and C2 spinal nerves, creating connections with motor regulatory pathways in the brainstem and basal ganglia. Pilot studies suggest that high-frequency stimulation of IAMZ can alleviate PD motor symptoms beyond the stimulation period.

This study aims to evaluate the safety and effectiveness of the EarStim System for intermittent symptom relief in PD patients. The study is a prospective, multi-center, randomized, two-period, non-significant risk pivotal study involving patients with PD experiencing wearing-off phenomena. It is designed to assess the safety and effectiveness of the EarStim System for the intermittent relief of motor symptoms. The study will recruit adult patients with moderate to severe PD, defined as an MDS-UPDRS Part III score of ≥33, who are being treated with oral dopaminergic medication.

The study consists of two periods: Period A and Period B. Period A will be a double-blind, randomized, sham-controlled part to assess the safety and effectiveness of the EarStim System in a clinical setting at Visit 1 (Day 0). Period B will be unblinded and controlled by a SOC arm to evaluate the effectiveness of the EarStim System in a home setting over a 90-day period.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling the following criteria are eligible for participation:

* Subject must be ≥44 years of age.
* Subject has PD and is on stable carbidopa/levodopa therapy for at least four weeks prior to enrollment in the study.
* Subject must be willing and able to refrain from changing PD medications or dosages during the 90-day study.
* Subject reports experiencing both "ON" and "OFF" episodes (MDS-UPDRS Part IV - Time Spent in the OFF-state score ≥1), as assessed and determined by the investigator.

  *This corresponds to item 4.3 in MDS-UPDRS Part IV, where a score of 0 (zero) indicates that the subject experiences no OFF periods during the waking day, and a score of ≥1 reflects the presence of OFF periods at any level.
* Subject experiences "OFF" periods with an "ON" score that is ≥20% better than the "OFF" score, as measured by the MDS-UPDRS Part III score, 1 hour after taking their dose of carbidopa/levodopa.
* Subject has an MDS-UPDRS Part III score ≥33 in "OFF" period.
* Subject agrees to remain in an "OFF" period for up to 3 hours without requiring rescue medication.
* Subject can walk independently, without the use of an assisted device (e.g., cane or walker), in both "ON" and "OFF" periods.
* Subject is willing to provide informed consent to participate in the study.
* Subject is willing and able to comply with all study procedures and required availability for study visits.

Exclusion Criteria:

Patients who meet any of the following criteria are to be excluded from participation:

* Subject has a medical or psychiatric comorbidity that may compromise participation in the study.
* Subject has a history of cardiac rhythm disorders (e.g., atrial fibrillation, ventricular tachycardia, or atrioventricular block).
* Subject is pregnant or planning to become pregnant during the course of the study.
* Subject has a form of Parkinsonism other than PD, such as drug-induced Parkinsonism or Multiple System Atrophy.
* Subject is currently using on-demand medications for PD, such as subcutaneous apomorphine, sublingual apomorphine, and levodopa inhalation powder.
* Subject has an implanted deep brain stimulator (DBS).
* Subject is receiving direct intestinal infusions of levodopa.
* Subject has a history of epilepsy.
* Subject's medications are expected to change during the 90-day study period.
* Subject has a cardiac pacemaker, defibrillator, bladder stimulator, spinal cord stimulator, or any other active electronic medical device.
* Subject is unable to understand or follow the instructions required by the study.
* Subject has an ear infection or skin condition around the ear.
* Subject is participating, or has participated, in another interventional clinical trial in the last 30 days that may confound the results of this study, unless approved by the Sponsor.
* Subject has a history of brain surgery or peripheral neuropathy.
* Subject is actively using TENS or has a history of chronic TENS use within the last 2 weeks prior to study enrollment.
* Subject consumed alcohol or caffeine within 12 hours of study enrollment or has a history of alcohol dependence

Min Age: 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in MDS-UPDRS III scores | 40 minutes
  Comparison of reduction in the MDS-UPDRS Part III scores from pre-stimulation to 40 minutes post-stimulation between active and sham arms during Period A.
Adverse events | From enrollment to the end of study at 90 days
  Frequency of all adverse events

SECONDARY OUTCOMES:
Change in MDS-UPDRS III score | 90 minutes
  Comparison of reduction in the MDS-UPDRS Part III scores from pre-stimulation to 90 minutes post-stimulation, comparing the active and sham arms during Period A (Visit 1).
Change in MDS-UPDRS III score | From 30 days (Visit 2) to 90 days (Visit 4)
  Mean reduction in the MDS-UPDRS Part III score from pre-stimulation to 40 minutes post-stimulation in the EarStim + SOC group compared with SOC group at Visit 2,3,4.
Change in MDS-UPDRS III score | 90 days
  Non-inferiority of the mean reduction in the MDS-UPDRS Part III score from pre-stimulation to 40 minutes post-stimulation in the EarStim + SOC group at Visit 4 compared with the active group at Visit 1.

OTHER OUTCOMES:
Patient Global Impression - Change (PGI-C) scale | 40 minutes
  Comparison of PGI-C scale scores between the active and sham arms after 40 minutes of stimulation at Visit 1.
Clinical Global Impression - Change (CGI-C) scale | 40 minutes
  Comparison of CGI-C scale scores between the active and sham arms after 40 minutes of stimulation at Visit 1.
Parkinson's Disease Questionnaire (PDQ-8) | From 30 days (Visit 2) to 90 days (Visit 4)
  Comparison of PDQ-8 scores between the "EarStim + SOC" and "SOC" groups at Visits 2, 3, and 4.
Parkinson's Disease Questionnaire (PDQ-8) | From Day -1 to 90 days (Visit 4)
  Comparison of PDQ-8 scores in the "EarStim + SOC" group at Visits 2, 3, and 4 versus the day before Visit 1.
MDS-UPDRS Part II scores | From Day 0 (Visit 1) to Day 90 (Visit 4)
  Comparison of the MDS-UPDRS Part II (Motor Aspects of Experiences of Daily Living) scores in the "EarStim + SOC" group between Visit 4 and Visit 1.
MDS-UPDRS Part I scores | From Day 0 (Visit 1) to Day 90 (Visit 4)
  Comparison of the MDS-UPDRS Part II (Non-Motor Aspects of Experiences of Daily Living) scores in the "EarStim + SOC" group between Visit 4 and Visit 1.
Parkinson's KinetiGraph (PKG™) | From baseline up to 90 days (Visit 4)
  Changes in PKG™ sleep and nighttime activity levels from pre-Visit 1 scores to the mean scores of Visits 2, 3, and 4.
Parkinson's KinetiGraph (PKG™) | From baseline up to 90 days (Visit 4)
  Changes in PKG™ motor fluctuations from pre-Visit 1 scores to the mean scores of Visits 2, 3, and 4.
Parkinson's KinetiGraph (PKG™) | From baseline up to 90 days (Visit 4)
  Changes in PKG™ bradykinesia, dyskinesia, and tremor from pre-Visit 1 scores to the mean scores of Visits 2, 3, and 4.
Wearing-off Questionnaire (WOQ-9) | From baseline up to 90 days (Visit 4)
  Comparison of Wearing-off Questionnaire (WOQ-9) scores between pre-Visit 1 and Visits 2, 3, and 4.
Change in MDS-UPDRS III score | 40 minutes
  Assessment of whether the mean reduction in the MDS-UPDRS Part III score from pre-stimulation to 40 minutes post-stimulation in the active arm at Visit 1 is clinically meaningful (≥3.2 points).
Change in MDS-UPDRS III score | 90 minutes
  Assessment of whether the mean reduction in the MDS-UPDRS Part III score from pre-stimulation to 90 minutes post-stimulation in the active arm at Visit 1 is clinically meaningful (≥3.2 points).
Change in MDS-UPDRS III score | From Day 0 (Visit 1) up to 90 days (Visit 4)
  Assessment of whether the mean reduction in the MDS-UPDRS Part III score from pre-stimulation to 40 minutes post-stimulation in "EarStim+SOC" group, combined across Visit 2,3,4 is clinically meaningful (≥3.2 points).

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Özgür Çakmak, MD, PhD, Assoc.Prof, Study Director — Stoparkinson Healthcare Systems LLC
Locations (2):
- Turkey (Türkiye) (2):
  - Koc University Hospital, Istanbul
  - Şişli Hamidiye Etfal Research and Training Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No